CLINICAL TRIAL: NCT02055365
Title: Effects of Persistent Innate Immune Activation on Vaccine Efficacy Pilot Study: Gene Expression Profiling of Immune Response to HBV Vaccination in Healthy Volunteers
Brief Title: Pilot Study: Gene Expression Profiling of Immune Response to HBV Vaccination in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Principal Investigator, Brad Rosenberg, Whitehead Presidential Fellow, Rockefeller University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BRO-0828
Record Dates: First submitted 2014-02-03; First posted 2014-02-05 (Estimated); Results first posted 2018-04-05 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-04

CONDITIONS: Hepatitis B
Keywords: Hepatitis B vaccine
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hepatitis B vaccination (Experimental): All subjects will receive the standard 3-dose course of Recombivax HB (Merck) - Hepatitis B Vaccine (Recombinant).
  Interventions: Biological: Hepatitis B Vaccine (Recombinant)

INTERVENTIONS:
Biological: Hepatitis B Vaccine (Recombinant) — All subjects will receive the standard 3-dose course of Recombivax HB (Merck) - Hepatitis B Vaccine (Recombinant).
  Other Names: Recombivax HB - Merck & Co., Inc.

SUMMARY:
Vaccines have been responsible for preventing millions of deaths and extending the average human lifespan. Effective vaccines stimulate the cells of the immune system to activate genes and associated functions that bring about protective immunity.This study aims to define cellular functions and genes important for the hepatitis B (HBV) vaccine immune response in healthy individuals. The investigators hypothesize that many genes associated with innate and adaptive immune functions are important for an effective HBV vaccine response.

DETAILED DESCRIPTION:
Vaccines have been responsible for preventing millions of deaths and extending the average human lifespan. Effective vaccines stimulate the cells of the immune system to activate genes and associated functions that bring about protective immunity. Knowledge of those genes and cellular functions activated by effective vaccination can improve our understanding of how the immune system works and define the features necessary for a successful vaccine response. This study aims to define cellular functions important for the hepatitis B (HBV) vaccine immune response in healthy individuals. The investigators will identify those genes that are activated or suppressed in immune cells at various times after each dose of the HBV vaccine. The investigators will explore these vaccine-induced "gene signatures" to characterize the cellular functions associated with an effective immune response to HBV vaccination. The investigators hypothesize that many genes associated with innate and adaptive immune functions are important for an effective HBV vaccine response.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer without significant medical problems
* Willing to receive three doses of an FDA-approved Hepatitis B vaccine

Exclusion Criteria:

* Male or female < 18 and > 60 years of age
* Received any vaccine within a month prior to study vaccine
* History of Hepatitis B infection
* History of previous Hepatitis B vaccination(s)
* History of Hepatitis C virus (HCV) infection or positive HCV antibody test
* Participation in another clinical study of an investigational product currently or within the past 90 days, or expected participation during this study
* Positive serum antibody against Hep B surface antigen and/or core Hep B core antigen
* human immunodeficiency virus (HIV) positive
* In the opinion of the investigator, the volunteer is unlikely to comply with the study protocol
* Any clinically significant abnormality or medical history or physical examination including history of immunodeficiency or autoimmune disease
* Is pregnant or lactating
* Currently taking systemic steroids or other immunomodulatory medications including anticancer medications and antiviral medications
* Any clinically significant acute or chronic medical condition requiring care by a primary care provider (e.g., diabetes, coronary artery disease, rheumatologic illness, malignancy, substance abuse) that, in the opinion of the investigator, would preclude participation
* Unable to continue participation for 30 weeks

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-02-18 (Actual); Primary Completion 2015-01-06 (Actual); Study Completion 2015-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brad Rosenberg, MD, PhD, Principal Investigator — The Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Hepatitis B Vaccination: All subjects will receive the standard 3-dose course of Recombivax Hepatitis B (HB) (Merck) - Hepatitis B Vaccine (Recombinant).
  Hepatitis B Vaccine (Recombinant): All subjects will receive the standard 3-dose course of Recombivax HB (Merck) - Hepatitis B Vaccine (Recombinant).
Period: Overall Study
Arm/Group | Hepatitis B Vaccination
Started | 10
Completed | 9
Not Completed | 1
Not completed — Prematurely Withdrawn | 1

BASELINE CHARACTERISTICS:
Arm/Group | Hepatitis B Vaccination
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Differentially Expressed Genes at p < 0.05 (Without Multiple Testing Correction).
Description: Number of differentially expressed genes at time point versus prevaccination baseline (p<0.05). Following Principal Components Analysis, data from one participant series was identified as a technical outlier and excluded from downstream analyses. Differential gene expression analysis was conducted with the voom/limma tools in the R statistical framework.
Time Frame: Day 1, Day 3, Week 1, and Week 2
Population: All participants received the standard 3-dose course of Recombivax HB (Merck) - Hepatitis B Vaccine (Recombinant). RNA-Seq (RNA sequencing) data from whole blood (PAXgene) for 9 participants were analyzed for differential gene expression at day 1, day 3, week 1, and week 2 after administration of the Hepatitis B Vaccine (Recombinant) (dose #1).
Measure: Number; unit: number of genes at p<0.05
Groups:
- Day 1: Differentially expressed genes at Day 1 versus pre-vaccination baseline (p<0.05).
- Day 3: Differentially expressed genes at Day 3 versus pre-vaccination baseline (p<0.05).
- Week 1: Differentially expressed genes at Week 1 versus pre-vaccination baseline (p<0.05).
- Week 2: Differentially expressed genes at Week 2 versus pre-vaccination baseline (p<0.05).
Arm/Group | Day 1 | Day 3 | Week 1 | Week 2
Number analyzed (Participants) | 9 | 9 | 9 | 9
number of genes at p<0.05
  Downregulated: number analyzed (Participants) | 8 | 8 | 8 | 8
  Downregulated | 138 | 138 | 102 | 81
  Unchanged: number analyzed (Participants) | 8 | 8 | 8 | 8
  Unchanged | 11139 | 11318 | 11189 | 11361
  Upregulated: number analyzed (Participants) | 8 | 8 | 8 | 8
  Upregulated | 316 | 137 | 302 | 151

2. Primary Outcome: Number of Significantly Differentially Expressed Genes at False Discovery Rate (FDR)< 0.05 (Upon Correction for Multiple Testing).
Description: Number of significantly differentially expressed genes at time point versus prevaccination baseline (FDR<0.05). Following Principal Components Analysis, data from one participant series was identified as a technical outlier and excluded from downstream analyses. Differential gene expression analysis was conducted with the voom/limma tools in the R statistical framework.
Time Frame: Day 1, Day 3, Week 1, and Week 2
Population: All participants received the standard 3-dose course of Recombivax HB (Merck) - Hepatitis B Vaccine (Recombinant). RNA-Seq data from whole blood (PAXgene) for 9 participants were analyzed for differential gene expression at day 1, day 3, week 1, and week 2 after administration of the Hepatitis B Vaccine (Recombinant) (dose #1).
Measure: Number; unit: number of genes at FDR<0.05
Groups:
- Day 1: Significantly Differentially expressed genes at Day 1 versus pre-vaccination baseline (FDR<0.05).
- Day 3: Significantly Differentially expressed genes at Day 3 versus pre-vaccination baseline (FDR<0.05).
- Week 1: Significantly Differentially expressed genes at Week 1 versus pre-vaccination baseline (FDR<0.05).
- Week 2: Significantly Differentially expressed genes at Week 2 versus pre-vaccination baseline (FDR<0.05).
Arm/Group | Day 1 | Day 3 | Week 1 | Week 2
Number analyzed (Participants) | 9 | 9 | 9 | 9
number of genes at FDR<0.05
  Downregulated: number analyzed (Participants) | 8 | 8 | 8 | 8
  Downregulated | 0 | 0 | 0 | 0
  Unchanged: number analyzed (Participants) | 8 | 8 | 8 | 8
  Unchanged | 0 | 0 | 0 | 0
  Upregulated: number analyzed (Participants) | 8 | 8 | 8 | 8
  Upregulated | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Hepatitis B Vaccination
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 2/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hepatitis B Vaccination (N=9)
Scratchy Throat (Respiratory, thoracic and mediastinal disorders) | 1
mild ecchymosis (Skin and subcutaneous tissue disorders) | 1
light headedness (Nervous system disorders) | 1

LIMITATIONS AND CAVEATS:
Although RNA-Seq analysis was effective in measuring gene expression levels, additional study subjects (more samples) may have improved statistical power to detect subtle changes in gene expression over time post-vaccination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes